CLINICAL TRIAL: NCT03775590
Title: The Role of Bathing Additives in the Treatment of Pediatric Atopic Dermatitis
Acronym: ASPIRE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed due to lack of enrollment.
Sponsor: Mayo Clinic (Other)
Collaborators: HealthPartners Institute (Other)
Responsible Party: Principal Investigator, Megha M. Tollefson, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18-006224
Record Dates: First submitted 2018-11-06; First posted 2018-12-14 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Atopic Dermatitis; Eczema
Keywords: Atopic Dermatitis; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — Water; Acetic Acid

STUDY DESIGN:
Intervention Model Description: There are 3 study arms with 50 subjects in each arm. The 3 arms are: water, water + bleach, and water + vinegar
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Water (Active Comparator): Subjects will bathe at least twice a week in a water bath for 6 months and keep a record of their bathing regimen
  Interventions: Procedure: Water
- Bleach (Active Comparator): Subjects will bathe at least twice a week in a water + dilute bleach bath for 6 months and keep a record of their bathing regimen
  Interventions: Procedure: Bleach
- Acetic acid (Active Comparator): Subjects will bathe at least twice a week in a water bath + vinegar for 6 months and keep a record of their bathing regimen
  Interventions: Procedure: Acetic acid

INTERVENTIONS:
Procedure: Water — To evaluate using water in the treatment of atopic dermatitis
  Arms: Water
Procedure: Bleach — To evaluate using water + dilute bleach in the treatment of atopic dermatitis
  Arms: Bleach
Procedure: Acetic acid — To evaluate using water + vinegar in the treatment of atopic dermatitis
  Other Names: vinegar
  Arms: Acetic acid

SUMMARY:
To evaluate the efficacy of water bath, water + bleach, and water + vinegar (acetic acid) in the treatment of atopic dermatitis (eczema)

DETAILED DESCRIPTION:
To perform a randomized controlled study to evaluate the efficacy of adding dilute acetic acid to the bath twice weekly on the Eczema Area and Severity Index (EASI) score as compared to adding dilute bleach to the bath including a control arm in which no solution is added to the bath.

ELIGIBILITY:
Inclusion Criteria:

* Currently reside in the USA
* Ability to comply with follow up visits at 2-4 months and at 6 months
* Come to the last follow-up at 6 months in the clinic
* At least 5% Body Surface Area (BSA) affected with AD

Exclusion Criteria:

* Unclear diagnosis of atopic dermatitis
* Inability to comply with additive baths
* Inability to comply with follow-up visits
* Lack of residence in the United States

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Eczema Area and Severity Index (EASI) score improvement from baseline | At each visit until the last visit at 6 months
  The EASI score is a validated composite score that ranges from 0 (clear) to 72 (very severe). The EASI is assessed and calculated as: the proportion of affected body surface area (BSA) was estimated from 4 designated body regions (head/neck, upper limbs, trunk, and lower limbs), and the Physician's Assessment of Individual Signs was determined for each region. The Physician's Assessment of Individual Signs grades signs of AD (erythema, edema/induration/papulation, excoriation, oozing/weeping/crusting, scaling, and lichenification) on a 4-point scale, ranging from absent to severe. Both the proportion of affected BSA and the Physician's Assessment of Individual Signs score are used to calculate the EASI score.

SECONDARY OUTCOMES:
Patient Oriented Eczema Measure (POEM) | At each visit until the last visit at 6 months
  The POEM measures the severity of eczema from a scale of 0-28 with 0 being clear and 28 as having severe eczema.
  * 0 to 2 = Clear or almost clear
  * 3 to 7 = Mild eczema
  * 8 to 16 = Moderate eczema
  * 17 to 24 = Severe eczema
  * 25 to 28 = Very severe eczema
Infant Dermatitis Quality of Life (IDQOL) for children under 4 years old | At each visit until the last visit at 6 months
  This quality of life (QoL) measures the patient quality of life from 0 - 30 with 0 being the patient's eczema doesn't have an affect on the patient's QoL while 30 means it has a profound effect on the patient's QoL.
Children's Dermatitis Quality of Life Index (CDQLI) for children at 4 years old or greater | At each visit until the last visit at 6 months
  This quality of life (QoL) measures the patient quality of life from 0 - 30 with 0 being the patient's eczema doesn't have an affect on the patient's QoL while 30 means it has a profound effect on the patient's QoL.
Rate of oral antibiotic prescribing | At each visit until the last visit at 6 months
  The number of oral courses of antibiotics given for skin related concerns at 2-4 months and at 6 months in each group.
Presence of staphylococcus aureus on involved skin | At each visit until the last visit at 6 months
  Differences in S. aureus colonization rates between each study arm at 2-4 months and at 6 months.
Changes in Investigator's Global Assessment (IGA) score from baseline | At each visit until the last visit at 6 months
  The IGA score (clear, almost clear, mild, moderate, severe, very severe; on numbered scaled where 0 = clear and 5 = very severe) at each visit
Frequency and severity of atopic dermatitis flares | At each visit until the last visit at 6 months
  Number and severity of flares in each group within 2-4 months and within 6 months
pH of the skin | At each visit until the last visit at 6 months
  Differences between the pH of the skin between the three study arms at 2-4 months and at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Megha M Tollefson, MD, Principal Investigator — Mayo Clinic; Sarah Asch, MD, Principal Investigator — HealthPartners Institute
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - HealthPartners, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eichenfield LF, Tom WL, Berger TG, Krol A, Paller AS, Schwarzenberger K, Bergman JN, Chamlin SL, Cohen DE, Cooper KD, Cordoro KM, Davis DM, Feldman SR, Hanifin JM, Margolis DJ, Silverman RA, Simpson EL, Williams HC, Elmets CA, Block J, Harrod CG, Smith Begolka W, Sidbury R. Guidelines of care for the management of atopic dermatitis: section 2. Management and treatment of atopic dermatitis with topical therapies. J Am Acad Dermatol. 2014 Jul;71(1):116-32. doi: 10.1016/j.jaad.2014.03.023. Epub 2014 May 9. PMID 24813302
- [Background] Huang JT, Abrams M, Tlougan B, Rademaker A, Paller AS. Treatment of Staphylococcus aureus colonization in atopic dermatitis decreases disease severity. Pediatrics. 2009 May;123(5):e808-14. doi: 10.1542/peds.2008-2217. PMID 19403473
- [Background] Hon KL, Tsang YC, Lee VW, Pong NH, Ha G, Lee ST, Chow CM, Leung TF. Efficacy of sodium hypochlorite (bleach) baths to reduce Staphylococcus aureus colonization in childhood onset moderate-to-severe eczema: A randomized, placebo-controlled cross-over trial. J Dermatolog Treat. 2016;27(2):156-62. doi: 10.3109/09546634.2015.1067669. Epub 2015 Aug 13. PMID 26270469
- [Background] Gonzalez ME, Schaffer JV, Orlow SJ, Gao Z, Li H, Alekseyenko AV, Blaser MJ. Cutaneous microbiome effects of fluticasone propionate cream and adjunctive bleach baths in childhood atopic dermatitis. J Am Acad Dermatol. 2016 Sep;75(3):481-493.e8. doi: 10.1016/j.jaad.2016.04.066. PMID 27543211
- [Background] Eichenfield LF, Tom WL, Chamlin SL, Feldman SR, Hanifin JM, Simpson EL, Berger TG, Bergman JN, Cohen DE, Cooper KD, Cordoro KM, Davis DM, Krol A, Margolis DJ, Paller AS, Schwarzenberger K, Silverman RA, Williams HC, Elmets CA, Block J, Harrod CG, Smith Begolka W, Sidbury R. Guidelines of care for the management of atopic dermatitis: section 1. Diagnosis and assessment of atopic dermatitis. J Am Acad Dermatol. 2014 Feb;70(2):338-51. doi: 10.1016/j.jaad.2013.10.010. Epub 2013 Nov 27. PMID 24290431
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials